CLINICAL TRIAL: NCT07083362
Title: Safety, Tolerability and Pharmacokinetic Studies of Single and Multiple Administrations of HRS-8829 in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Study of HRS-8829
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-8829-101
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemia Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group 1 (Experimental)
  Interventions: Drug: HRS-8829;Placebo
- Treatment group 2 (Experimental)
  Interventions: Drug: HRS-8829;Placebo
- Treatment group 3 (Experimental)
  Interventions: Drug: HRS-8829;Placebo
- Treatment group 4 (Experimental)
  Interventions: Drug: HRS-8829;Placebo

INTERVENTIONS:
Drug: HRS-8829;Placebo — Subject will receive HRS-8829 at dose level 1.
  Subject will receive placebo at dose level 1.
  Arms: Treatment group 1
Drug: HRS-8829;Placebo — Subject will receive HRS-8829 at dose level 2.
  Subject will receive placebo at dose level 2.
  Arms: Treatment group 2
Drug: HRS-8829;Placebo — Subject will receive HRS-8829 at dose level 3.
  Subject will receive placebo at dose level 3.
  Arms: Treatment group 3
Drug: HRS-8829;Placebo — Subject will receive HRS-8829 at dose level 4.
  Subject will receive placebo at dose level 4.
  Arms: Treatment group 4

SUMMARY:
This study adopted a single-center, randomized, double-blind, placebo-controlled, dose-escalation design and was divided into two parts: single-dose dose-escalation (SAD) and multiple-dose dose-escalation (MAD)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 55 years old
2. The weight of female subjects was ≥45 kg, that of male subjects was ≥50 kg, and the body mass index (BMI) was within the range of 19.0-28.0 kg/m2
3. The female subjects were not in the pregnancy or lactation period, and the pregnancy examination results before the test were negative; Male or female subjects agreed to take the investigator-approved effective contraceptive measures during the trial as required by the investigator.
4. Voluntarily participate in this clinical trial

Exclusion Criteria:

1. Have any history of allergies
2. Have had or are currently suffering from diseases of the heart, liver, kidneys, endocrine system, digestive tract, immune system, respiratory system, musculoskeletal system and nervous system, etc
3. The electrocardiogram at lead 12 was abnormal and was judged by the researcher as unsuitable to participate in this study
4. Those who test positive for any one of hepatitis B surface antigen, hepatitis C antibody, syphilis specific antibody or human immunodeficiency virus antigen-antibody during the screening period
5. Those whose screening period examination results are judged by the research doctor as abnormal and of clinical significance
6. Those who have used any drugs that inhibit or induce liver enzymes within one month before administration
7. Those who have used or are currently using any medication within two weeks prior to administration
8. Those who have received a vaccine within one month prior to screening (except for the influenza vaccine) or plan to receive a vaccine during the trial period
9. Those who have undergone major surgical operations within the six months prior to screening
10. Blood donation or loss of more than 400 mL within 3 months prior to screening
11. Participate in the clinical trial of the drug as a subject and take the trial drug
12. Consumed more than 14 units of alcohol per week on average within the 3 months prior to screening
13. Those who smoked more than 5 cigarettes or an equivalent amount of tobacco per day
14. Those who consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice and/or caffeinated beverages daily
15. Consume special food within 48 hours before administration
16. Those with a history of drug abuse
17. Those who cannot tolerate venipuncture
18. Those who have special dietary requirements
19. The researchers believe that the subjects have any other factors that make them unsuitable for participating in this trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | From ICF signing date to Day8 after single administration
The incidence and severity of adverse events | From ICF signing date to Day15 after multiple administrations

SECONDARY OUTCOMES:
Maximum observed concentration of HRS-8829 and its metabolite in plasma (Cmax) | 0 hour to 48 hour after single administration
Area under the serum concentration time curve (AUC) of HRS-8829 and its metabolite in plasma | 0 hour to 48 hour after single administration
Time to maximum observed concentration (Tmax) of HRS-8829 and its metabolite in plasma | 0 hour to 48 hour after single administration
Half-life (T1/2) of HRS-8829 and its metabolite in plasma | 0 hour to 48 hour after single administration
Clearance (CL) of HRS-8829 and its metabolite in plasma | 0 hour to 48 hour after single administration
Volume of distribution (Vz) of HRS-8829 and its metabolite in plasma | 0 hour to 48 hour after single administration
Cumulative amount excreted (Ae0-t) of HRS-8829 and its metabolite in urine | 0 hour to 48 hour after single administration
Cumulative excretion fraction (Fe0-t) of HRS-8829 and its metabolite in urine | 0 hour to 48 hour after single administration
Renal clearance (CLr) of HRS-8829 and its metabolite in urine | 0 hour to 48 hour after single administration
Maximum observed concentration at steady-state of HRS-8829 and its metabolite in plasma (Cmax) | Day1 to Day15 after multiple administrations
Area under the serum concentration time curve (AUC) at steady-state of HRS-8829 and its metabolite in plasma | Day1 to Day15 after multiple administrations
Time to maximum observed concentration (Tmax) of HRS-8829 and its metabolite in plasma | Day1 to Day15 after multiple administrations
Half-life (T1/2) of HRS-8829 and its metabolite in plasma | Day1 to Day15 after multiple administrations
Clearance (CL) of HRS-8829 and its metabolite in plasma | Day1 to Day15 after multiple administrations
Volume of distribution (Vz) of HRS-8829 and its metabolite in plasm | Day1 to Day15 after multiple administrations

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided